CLINICAL TRIAL: NCT05841953
Title: The Use of Electrical Stimulation to Increase Anal Pressures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dan Livovsky, Director of Neurogastroenterology, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0020-23-SZMC; MOH_2023-04-16_012540 (Registry Identifier: Israel Ministry of Healt Clinical Trials Registry (in Hebrew))
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single arm (Experimental): All participant will be exposed to the full stimulation protocol 2 different protocols using 2 different electrode arrays will be studied in random order.
  Interventions: Device: Transcutaneous neuromuscular electrical stimulation

INTERVENTIONS:
Device: Transcutaneous neuromuscular electrical stimulation — Transcutaneous electrical stimulation will be delivered to the anal sphincter and anal resting and squeezing pressures as a result of the stimulation will be recorded for different stimulation protocols using approved electrotherapy units

SUMMARY:
The goal of this clinical trial is to learn about the feasibility of inducing contraction of the anal sphincter by transcutaneous neuromuscular electrical stimulation in patients with fecal incontinence.

The main questions it aims to answer are:

* Efficacy of the specific stimulation protocol to increase anal pressures
* Tolerability and safety Participants will be exposed to the stimulation with the changes in pressure will be studied using high resolution anorectal manometry

ELIGIBILITY:
Inclusion Criteria:

* Undergoing anorectal manometry for the evaluation of fecal incontinence indication
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* >18 years old

Exclusion Criteria:

* Pregnant or attempting to become pregnant. The safety of electronic muscle stimulators during pregnancy has not been established.
* An electronic implant (e.g. cardiac pacemaker, implanted defibrillator) or suffer from heart problems.
* Conductive intra-uterine devices (IUD/Coil) or metal implants in the abdominal or pelvic area, including the hip and lumbar spine
* Cancer, epilepsy, or cognitive dysfunction.
* Pelvic floor surgery within the last six weeks.
* Complete denervation of the pelvic floor.
* Advanced full thickness rectal prolapse.
* Injured, inflamed or any significant disease in the peri-anal skin.
* Allergy to any component of the device, either known of developed during testing.
* Moderate to severe proctitis of any etiology.
* Skin irritation at the site of the stimulating electrodes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Stimulation intensity levels | During exposure to electrical stimulation 5 min
  The stimulation intensity levels measured in milliamperes (mA) required to induce changes in anal sphincter pressures measured by manometry.

SECONDARY OUTCOMES:
Maximal tolerability to neuromuscular transcutaneous stimulation measured as the current in mA causing discomfort of at least 7 on a scale of 0 to 10 points. | During exposure to electrical stimulation 5 min
  The stimulation intensity levels measured as the current in milliamperes (mA) causing a discomfort level of 7 out of 10 point or the current at which a participant asks to stop the stimulation.
Safety of neuromuscular transcutaneous stimulation measured as the proportion of patients reporting or presenting with adverse events during the study attributed or not to the use of electrical stimulation | Until discharge, assessed up to 7 days
  The Rate of Adverse Events (e.g., pain, skin reactions, prolonged abnormal sensation after stopping the stimulation, etc.) during the study attributed or not to the use of electrical stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Diseases Institute, Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
Data will not be anonymized; thus, due to privacy rights, we will consider the ethical and legal implications of sharing the data, providing that a relevant request for data is received.

REFERENCES:
- [Background] Livovsky DM, Koslowsky B, Goldin E, Lysy J. External kinesiology tape for improvement in fecal incontinence symptom bother in women: a pilot study. Int Urogynecol J. 2022 Oct;33(10):2859-2868. doi: 10.1007/s00192-021-05050-z. Epub 2022 Jan 18. PMID 35039916
- [Background] Riedy LW, Chintam R, Walter JS. Use of a neuromuscular stimulator to increase anal sphincter pressure. Spinal Cord. 2000 Dec;38(12):724-7. doi: 10.1038/sj.sc.3101088. PMID 11175371